CLINICAL TRIAL: NCT02934932
Title: A Pilot Dose-Response Biomarker Study of Brexpiprazole Treatment in PTSD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to slow enrollment.
Sponsor: Duke University (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00071923
Record Dates: First submitted 2016-10-14; First posted 2016-10-17 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — brexpiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Brexpiprazole 2mg (Experimental): Subjects will be titrated to this dose of brexpiprazole for 6 weeks.
  Interventions: Drug: Brexpiprazole
- Brexpiprazole 4mg (Experimental): Subjects will be titrated to this dose of brexpiprazole for 6 weeks.
  Interventions: Drug: Brexpiprazole
- Placebo (Placebo Comparator): Subjects will be titrated to this dose of placebo for 6 weeks.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Comparison of brexpiprazole 2mg to placebo Comparison of brexpiprazole 4mg to placebo
  Other Names: Rexulti

SUMMARY:
Determine if brexpiprazole treatment will be associated with a dose-dependent reduction in resting pupil diameter as a reflection of locus coeruleus (LC) norepinephrine (NE) neuron target engagement in a group of subjects with PTSD. All subjects will be evaluated by physical examination, ECG, standard blood chemistry, hematologic labs, toxicology testing, and urinalysis. Results of these studies must demonstrate a lack of clinically significant abnormalities prior to enrollment. Subjects will need to satisfy DSM-5 criteria for PTSD and receive a CAPS-5 score of 40 or greater on testing for study enrollment. Resting pupil diameter during pupillometric evaluation after two weeks on each treatment will serve as the primary outcome measure. This will be compared in the treatment groups using mixed effects repeated measures models to evaluate if there is a significant difference in pupil size among the treatments studied. As a secondary analysis this approach will be used to evaluate whether there is treatment effect on total CAPS-5 score. Lastly, the investigators will compute correlations between pupil size and CAPS-5 scores.

DETAILED DESCRIPTION:
Primary Hypothesis: Brexpiprazole treatment will be associated with dose-dependent reduction in resting pupil diameter as a reflection of LC NE neuron target engagement in a group of subjects with PTSD. Secondary Hypothesis: Brexpiprazole therapy will be associated with a dosedependent decrease in CAPS-5 scores Tertiary Hypothesis: The pre-post treatment change in resting pupil diameter will be statistically significantly correlated with the pre-post change in CAPS-5 score.

Subjects will be screened and will undergo pupil measures with rating scales on Visit 1. Subject must be free of all psychotropic medications for one week before Day 1 assessment, except that prior FLX treatment will require 4 weeks of abstinence, and MAOIs will require 2 weeks of abstinence. They will be randomized to study drug an issued six weeks of study medication on Day 1 to take home. A phone call will then occur for safety assessment and medication adherence at every week. They will present back to the study site on Day 42 and undergo pupil measures with rating scales. They will then undergo a one week washout period. On Day 49 they will then be given another study drug to take home with rating scales and pupil measures obtained that day. A phone call will then occur for safety assessment and medication adherence at every week. They will present back to the study site on Day 91 and undergo pupil measures with rating scales. They will then undergo a one week washout period. On Day 98 they will then be given another study drug to take home with rating scales and pupil measures obtained that day. A phone call will then occur for safety assessment and medication adherence at every week. They will present back to the study site on Day 140 and undergo pupil measures with rating scales. No more study medication will be provide on Day 140 and a final visit will be scheduled for on Day 147, one week later, for and end of study interview with labs and physical exam. At each visit, other than the final visit, subjects will complete the CAPS-5, MADRS, Insomnia Severity Index, and Clinician Assessment for Adverse Effects.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be 18-65 years of age.
* All subjects will be evaluated by physical examination, ECG, standard blood chemistry, hematologic labs, toxicology testing, and urinalysis at baseline and end of study. Results of these studies must demonstrate a lack of clinically significant abnormalities prior to enrollment. If results are outside of the normal reference range the study physician will be consulted to assess if clinically significant.
* Subjects will need to satisfy DSM-5 criteria for PTSD and receive a CAPS-5 score of 40 or greater on testing for study enrollment.
* Subjects will need to be free of psychotropic medications or treatments that could impact results of this study as deemed by the PI for at least 1 week.
* If the subject's primary psychiatrist or treating primary care physician are providing the subject with psychotropic medications they will be notified and a discussion about tapering current psychotropic medications prior to study enrollment will occur.

Exclusion Criteria:

1. Subjects will be excluded if they have significant medical or neurologic conditions (other than mild to moderate TBI), specifically seizures, or movement disorders,
2. have substance abuse within 12 months of study enrollment, substance dependence within past three months, per DSM-5 criteria (excluding caffeine and nicotine). The absence of substance use will be determined by self-report and confirmed by the results of urine toxicology at screening.
3. Women who are pregnant, breast-feeding, or planning to become pregnant while enrolled in this study will also be excluded.
4. Subjects with a history of severe drug allergy or hypersensitivity, or known hypersensitivity to the Brexpiprazole or its ingredients.
5. The subject has a history of tardive dyskinesia.
6. The subject has clinically significant extrapyramidal symptoms (EPS) including akathisia.
7. The subject has epilepsy or a history of seizures, except for a single seizure episode (e.g., childhood febrile seizure, post traumatic, or alcohol withdrawal).
8. The subject has chronic, uncontrolled, or unstable clinically relevant medical conditions Including:

   * Uncontrolled hypertension defined as blood pressure greater than 180/90
   * Hypotension defined as a blood pressure less than 90/60
   * Moderate to severe hepatic impairment (Child-Pugh score ≥7)
   * Moderate, Severe or End-Stage Renal Impairment (CrCL <60ml/min)
   * Known CYP2DG Poor Metabolizers
   * Heart failure NYHA Class III or IV
   * Diabetes mellitus or HbA1c greater than 5.7% (which defines pre-diabetes)
   * Hypertriglyceridemia defined as triglycerides greater than 200mg/dL
   * Low white blood cell count (below lower range of normal)
   * History of leukopenia or neutropenia
   * Arrhythmia with heart rate greater than 100bpm
   * Myocardial infarction in the past 6 months
   * Cerebrovascular accident in the past 6 months
   * Recurrent syncope
   * Seizure disorder
   * Currently receiving treatment for malignancy
   * QTc interval of greater than 450ms on electrocardiogram
9. The subject has a neurodegenerative disorder (Alzheimer disease, Parkinson's disease, multiple sclerosis, Huntington disease, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-25 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven T Szabo, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Pamela Smith, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 participants signed consent; 6 screen failed. All subjects received all three treatments with treatment order randomized within each subject.
Groups:
- All Participants: All participants who began the study.
Period: Overall Study
Arm/Group | All Participants
Started | 9
Completed | 6
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Six participants screen failed. All other subjects received all three treatments with treatment order randomized within each subject.
Groups:
- All Participants: All participants who signed consent.
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in Resting Pupil Diameter
Description: Evaluate the effects of two doses of brexpiprazole on locus coeruleus (LC) norepinephrine (NE) neuron activity.
Time Frame: Baseline to 6 weeks for each treatment arm
Population: Data not collected.
Groups:
- Brexpiprazole 2mg; Brexpiprazole 4mg: Subjects will be titrated to this dose of brexpiprazole for 6 weeks.
  Brexpiprazole: Comparison of brexpiprazole to placebo
- Placebo: Subjects will be titrated to this dose of placebo for 6 weeks.
  Brexpiprazole: Comparison of brexpiprazole to placebo
Arm/Group | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Change in CAPS-5 Ratings Score
Description: Determine the effect of brexpiprazole therapy on PTSD symptom severity
Time Frame: Baseline to 6 weeks for each treatment arm
Population: Data not collected.
Arm/Group | Brexpiprazole 2mg | Brexpiprazole 4mg | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT02934932/Prot_SAP_000.pdf